CLINICAL TRIAL: NCT03035344
Title: Study of the Intermediate Metabolism in Children With Acute Lymphoblastic Leukemia
Brief Title: Study of the Intermediate Metabolism in Children With Acute Lymphoblastic Leukemia (ALL)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Maria T. Papadopoulou, Principal investigator, MD, PhD candidate, Aristotle University Of Thessaloniki
Other Study IDs: CHILDHOOD ALL METABOLOMICS
Record Dates: First submitted 2017-01-26; First posted 2017-01-30 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric; Metabolism Disorder
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, bone marrow
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ALL paediatric patients: Metabolome study in children diagnosed with ALL after bone marrow biopsy
  Interventions: Other: Metabolome study
- Healthy matched controls: Metabolome study in healthy children matched for gender and age with the patients group
  Interventions: Other: Metabolome study

INTERVENTIONS:
Other: Metabolome study — Metabolome study in ALL patients compared to healthy controls

SUMMARY:
Study of the intermediate metabolism in children diagnosed with ALL compared to healthy matched controls.

DETAILED DESCRIPTION:
The primary cause of this study is to investigate the changes that ALL may cause to the metabolome of pediatric patients, in order to better understand its mechanism of action and target metabolic pathways for potential therapies.

ELIGIBILITY:
* Sex: all
* Minimum age: 1 year
* Maximum age: 16 years
* The study accepts healthy volunteers as matched controls for the patinets.
* Inclusion criteria: 1)Children diagnosed with ALL 2) Diagnosis confirmed with bone marrow biopsy 3) Sampling before the initiation of therapy 4) Informed consent signed
* Exclusion Criteria: 1) Children with a known chronic illness before ALL diagnosis 2) ALL remission 3) Not signed informed consent
* Population description: Patients are recruited from the Pediatric Hematology/Oncology Department of Aristotle University of Thessaloniki (AHEPA hospital) and from the Pediatric Hematology/ Oncology Department of Ippokration Hospital, that host all children diagnosed with ALL in nothern Greece. Matched controls are recruited from outpatient clinic of the 2nd and 4th Pediatric Department of Aristotle University of Thessaloniki.
* Sampling method: Non-probability sample

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children diagnosed with acute lymphoblastic leukemia
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Difference in measurement of aminoacids and organic acids between ALL patients and healthy matched controls. | Up to six months
  The title of aminoacids in blood and urine and of organic acids in urine will be measured through Tandem Mass Spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Athanassios Evangeliou, Prof, Study Chair — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided